CLINICAL TRIAL: NCT05063994
Title: A Randomized, Double-Blind, Active-Controlled, Phase 3 Study of Chronocort Compared With Immediate-Release Hydrocortisone Replacement Therapy in Participants Aged 16 Years and Over With Congenital Adrenal Hyperplasia
Brief Title: Comparison of Chronocort Versus Standard Hydrocortisone Replacement Therapy in Participants Aged 16 Years and Over With Congenital Adrenal Hyperplasia
Acronym: CONnECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIUR-014
Record Dates: First submitted 2021-05-28; First posted 2021-10-01 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chronocort (Experimental): Participants received Chronocort at a starting dose of 30 milligrams (mg), with dose adjustments down to 25, 20, or 15 mg based on adrenal insufficiency symptoms and androgen levels. Placebo was used for dose adjustment to maintain blinding.
  Interventions: Drug: Chronocort; Other: Placebo
- Cortef (Active Comparator): Participants received Cortef at a starting dose of 30 mg, with dose adjustments down to 25, 20, or 15 mg based on adrenal insufficiency symptoms and androgen levels. Placebo was used for dose adjustment to maintain blinding.
  Interventions: Drug: Cortef; Other: Placebo

INTERVENTIONS:
Drug: Chronocort — Over-encapsulated hydrocortisone modified-release capsule for oral administration.
  Other Names: Hydrocortisone modified-release
  Arms: Chronocort
Drug: Cortef — Over-encapsulated hydrocortisone immediate-release tablet for oral administration.
  Other Names: Immediate-release hydrocortisone; IRHC
  Arms: Cortef
Other: Placebo — Matching placebo

SUMMARY:
This study is a randomized, double-blind, active-controlled, phase III study of Chronocort® compared with immediate-release hydrocortisone replacement therapy in participants aged 16 years and over with Congenital Adrenal Hyperplasia.

DETAILED DESCRIPTION:
The study will compare the efficacy, safety and tolerability of twice daily Chronocort with twice daily immediate release hydrocortisone replacement therapy (IRHC) (Cortef®) in participants aged 16 years and over with known classic Congenital Adrenal Hyperplasia (CAH) due to 21 hydroxylase deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be aged 16 years or older at the time of signing the informed consent/assent.
* In participants aged <18 years, height velocity must be less than 2 cm/year in the last year and puberty must be completed (Tanner stage V).
* Participants with known classic CAH due to 21 hydroxylase deficiency diagnosed in childhood with documented (at any time) elevated 17-OHP and with or without elevated A4 and currently treated with hydrocortisone, prednisone, prednisolone or dexamethasone (or a combination of the aforementioned glucocorticoids) and on stable glucocorticoid therapy for a minimum of 3 months.
* Participants who are receiving fludrocortisone must be on a documented stable dose for a minimum of 3 months prior to enrollment and must have stable renin levels at screening.
* Female participants of childbearing potential and all male participants must agree to the use of an accepted method of contraception during the study.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and she is either not a woman of childbearing potential (WOCBP) or has a negative pregnancy test at entry into the study. Note: females presenting with oligomenorrhea or amenorrhea who are aged ≤55 years should be considered potentially fertile and therefore should undergo pregnancy testing like all other female participants.
* Capable of giving signed informed consent/assent which includes compliance with requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Clinical or biochemical evidence of hepatic or renal disease e.g. creatinine >2 times the upper limit of normal (ULN) or elevated liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2 times the ULN).
* History of bilateral adrenalectomy.
* History of malignancy (other than basal cell carcinoma successfully treated >26 weeks prior to entry into the study).
* Participants who have type 1 diabetes or receive regular insulin, have uncontrolled diabetes, or have a screening HbA1c greater than 8%.
* Persistent signs of adrenal insufficiency or the participant does not tolerate treatment at the end of the 4-week run-in period.
* Participants with any other significant medical or psychiatric conditions that in the opinion of the Investigator would preclude participation in the study.
* Participants on regular daily inhaled, topical, nasal or oral steroids for any indication other than CAH.
* Co-morbid condition requiring daily administration of a medication or consumption of any material that interferes with the metabolism of glucocorticoids.
* Participants who are receiving <10 mg hydrocortisone dose at screening or the hydrocortisone dose equivalent.
* Participants anticipating regular prophylactic use of additional steroids e.g. for strenuous exercise.
* Participation in another clinical study of an investigational or licensed drug or device within the 12 weeks prior to screening.
* Inclusion in any natural history or translational research study that would require evaluation of androgen levels during the study period outside of this protocol's assessments.
* Participants who have previously been exposed to Chronocort in any Diurnal study.
* Participants who routinely work night shifts and so do not sleep during the usual night-time hours.
* Participants, who in the opinion of the Investigator, will be unable to comply with the requirements of the protocol.
* Participants with a known hypersensitivity to any of the components of the Chronocort capsules, the Cortef tablets, or the placebo capsules.
* Participants with congenital galactosemia, malabsorption of glucose and galactose, or who are lactase deficient.
* Participants with a body weight of 45 kg or less.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Neurocrine UK Limited
Locations (21):
- United States (11):
  - Diurnal Investigational Site in Los Angeles, Los Angeles, California
  - Diurnal Investigational Site in Orange, Orange, California
  - Diurnal Investigational Site in Jacksonville, Jacksonville, Florida
  - Diurnal Investigational Site in Iowa, Iowa City, Iowa
  - Diurnal Investigational Site in Maryland, Bethesda, Maryland
  - Diurnal Investigational Site in Michigan, Ann Arbor, Michigan
  - Diurnal Investigational Site in Rochester, Rochester, Minnesota
  - Diurnal Investigational Site in Nevada, Las Vegas, Nevada
  - Diurnal Investigational Site in Dallas, Dallas, Texas
  - Diurnal Investigational Site in Seattle, Seattle, Washington
  - Diurnal Investigational Site in Milwaukee, Milwaukee, Wisconsin
- France (6):
  - Diurnal Investigational Site in Caen, Caen, Normandy
  - Diurnal Investigational Site in Pessac, Bordeaux
  - Diurnal Investigational Site in Bron, Lyon
  - Diurnal Investigational Site in Paris, Paris
  - Diurnal Investigational Site in Toulouse (Children's Hospital), Toulouse
  - Diurnal Investigational Site in Toulouse, Toulouse
- Japan (4):
  - Diurnal Investigational Site in Asahi-ku, Yokohama, Kanagawa
  - Diurnal Investigational Site in Yushima, Bunkyō-Ku, Tokyo
  - Diurnal Investigational Site in Okura, Setagaya-Ku, Tokyo
  - Diurnal Investigational Site in Toyama, Shinjuku-Ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received immediate-release hydrocortisone (IRHC; Cortef) during the run-in therapy for 4 weeks prior to randomization. Once eligibility for the study was confirmed at the Baseline visit, participants were randomized on a 1:1 basis (Chronocort:Cortef). 55 participants entered the run-in period and 53 were randomized to treatment.
Groups:
- Cortef Run-In: Participants received Cortef 30 milligrams (mg) total daily dose during the run-in therapy for 4 weeks prior to randomization.
- Chronocort: Participants received Chronocort at a starting dose of 30 mg, with dose adjustments down to 25, 20, or 15 mg based on adrenal insufficiency symptoms and androgen levels. Placebo was used for dose adjustment to maintain blinding.
Period: Cortef Run-In
Arm/Group | Cortef Run-In | Chronocort | Cortef
Started | 55 | 0 | 0
Completed | 53 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 0
Not completed — Did not meet the inclusion/exclusion criteria at end of Run-In | 1 | 0 | 0
Period: Treatment
Arm/Group | Cortef Run-In | Chronocort | Cortef
Started | 0 | 25 | 28
Full Analysis Set (FAS) Population (All participants with congenital adrenal hyperplasia (CAH) who were randomized into the study and who received at least 1 dose of study drug.) | 0 | 25 | 28
Completed | 0 | 25 | 25
Not Completed | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: FAS: All participants with congenital adrenal hyperplasia (CAH) who were randomized into the study and who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronocort | Cortef | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (14.68) | 31.6 (13.02) | 34.0 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 12 | 25
  Black or African American | 1 | 2 | 3
  Asian | 4 | 5 | 9
  Not Reportable | 6 | 6 | 12
  Unknown | 1 | 3 | 4
17-Hydroxyprogesterone (17-OHP) Level [Mean (Full Range); unit: nanograms (ng)/deciliters (dL)] | 3470.48 [43.5 to 16968.5] | 5595.36 [10.0 to 14641.5] | 4593.06 [10.0 to 16968.5]
Androstenedione (A4) Level [Mean (Full Range); unit: ng/dL] — Population: Participants in the FAS population who had an A4 assessment at the baseline visit.
  ng/dL
    number analyzed (Participants) | 25 | 27 | 52
    (all) | 173.30 [5.0 to 1040.5] | 483.09 [5.0 to 2516.5] | 334.15 [5.0 to 2516.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Biochemical Responders at Week 28
Description: Biochemical response was defined as a participant who a) was in biochemical control at the 08:00 assessment and b) was receiving a total daily dose of hydrocortisone of not more than 25 mg if the participant was in biochemical control at baseline or not more than 30 mg if the participant was not in biochemical control at baseline.
  Biochemical control was defined as both a 17-OHP concentration equal to or below the upper limit for optimal control (1200 ng/dL [36.4 nmol/L]) and an A4 concentration equal to or below the upper limit of the reference range (150 ng/dL [5.2 nmol/L] for men and 200 ng/dL [7.0 nmol/L] for women).
  Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 28
percentage of participants | 40.0 | 14.3
Statistical Analysis 1: Comparison: Chronocort vs Cortef; Test type: Non-Inferiority — Non-inferiority of Chronocort to Cortef was declared if the 95% CI for the difference in biochemical response rates between the 2 treatment arms (Chronocort minus Cortef) was wholly above minus 15 percentage points; p = 0.0003, Regression, Logistic — One-sided non-inferiority. The Ge et al (2011) method was used to calculate the estimate, standard error, confidence interval and P-value for the treatment difference from the results of a logistic regression analysis; Treatment Difference = 25.7, 95% CI 2-sided [2.5 to 48.9], Standard Error of Mean 11.82

2. Secondary Outcome: Percentage of Participants Who Were Dose Responders at Week 28
Description: Dose response was defined as a participant who a) was receiving a total daily dose of hydrocortisone of not more than 25 mg and b) was in biochemical control at the 08:00 assessment.
  Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 28
percentage of participants | 36.0 | 10.7
Statistical Analysis 1: Comparison: Chronocort vs Cortef; Test type: Superiority — Superiority of Chronocort to Cortef with respect to the dose response after 28 weeks of randomized treatment was declared if the two-sided 95% CI for the difference in response rates between the 2 treatment arms (Chronocort minus Cortef) was wholly above zero, provided that non-inferiority of Chronocort to Cortef with respect to the biochemical response had been declared under the primary efficacy objective; p = 0.012, Regression, Logistic — One-sided superiority. The Ge et al (2011) method was used to calculate the estimate, standard error, confidence interval and P-value for the treatment difference from the results of a logistic regression analysis; Treatment Difference = 25.3, 95% CI 2-sided [3.3 to 47.3], Standard Error of Mean 11.24

3. Secondary Outcome: Total Daily Dose of Hydrocortisone at Week 28
Description: Least squares (LS) mean was assessed using mixed model repeated measures (MMRM).
  Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 28
mg | 20.2 [17.8 to 22.6] | 26.0 [23.7 to 28.3]
Statistical Analysis 1: Comparison: Chronocort vs Cortef; Test type: Superiority — Superiority of Chronocort to Cortef (with respect to the total daily dose after 28 weeks of randomized treatment) was declared if the two-sided 95% CI for the difference in means between the 2 treatment arms (Chronocort minus Cortef) was wholly below zero, provided that non-inferiority of Chronocort to Cortef in terms of biochemical response had been declared under the primary efficacy objective, and superiority of Chronocort to Cortef in terms of dose response has been declared; p = 0.0005, MMRM — One-sided superiority; Treatment Difference = -5.8, 95% CI 2-sided [-9.2 to -2.5], Standard Error of Mean 1.66

4. Secondary Outcome: Number of Participants in Biochemical Control
Description: Biochemical control was defined as both a 17-OHP concentration (assessed at 08:00) equal to or below the upper limit for optimal control (1200 ng/dL [36.4 nmol/L]) and an A4 concentration equal to or below the upper limit of the reference range (150 ng/dL [5.2 nmol/L] for men and 200 ng/dL [7.0 nmol/L] for women).
  Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline and Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug. Participants with evaluable data for the endpoint were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Cortef: Participants received Chronocort at a starting dose of 30 mg, with dose adjustments down to 25, 20, or 15 mg based on adrenal insufficiency symptoms and androgen levels. Placebo was used for dose adjustment to maintain blinding.
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 27
Participants
  Baseline | 13 | 8
  Week 28: number analyzed (Participants) | 25 | 25
  Week 28 | 10 | 4

5. Secondary Outcome: Change From Baseline in Mean of 08:00 and 13:00 17-OHP Levels at Week 28
Description: LS mean was assessed using analysis of covariance (ANCOVA). Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline, Week 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 25
ng/dL | -1223.91 [-2897.42 to 449.6] | 1612.17 [-61.34 to 3285.68]

6. Secondary Outcome: Change From Baseline in Mean of 08:00 and 13:00 A4 Levels at Week 28
Description: LS mean was assessed using ANCOVA. Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline, Week 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 25
ng/dL | -4.85 [-115.57 to 105.86] | 146.13 [35.42 to 256.85]

7. Secondary Outcome: Number of Participants With Menstrual Regularity (Females of Childbearing Potential Only) at Week 28
Description: Data are presented for the number of participants with more than monthly menstrual cycles, monthly menstrual cycles, and number of participants with oligomenorrhoea and amenorrhoea. Oligomenorrhoea was defined as fewer than 9 menstrual cycles per year or cycle length >35 days and amenorrhoea as absent menses for ≥ 3 months.
  Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug. Only female participants of childbearing potential with evaluable data for the endpoint were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 14 | 12
Participants
  More than Monthly | 0 | 0
  Monthly | 9 | 2
  Oligomenorrhoea | 2 | 4
  Amenorrhoea | 3 | 6

8. Secondary Outcome: Change From Baseline in Luteinizing Hormone Levels (Males Only) at Week 28
Description: as for outcome 6
Time Frame: Baseline, Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug. Only male participants with evaluable data for the endpoint were analyzed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 9 | 10
mIU/mL | 0.15 [-0.71 to 1.02] | -1.19 [-2.01 to -0.37]

9. Secondary Outcome: Percent Change From Baseline in Size of Testicular Adrenal Rest Tumors at Week 28 (Males Only)
Description: Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Week 28
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 4 | 5
percent change | -7.67 (9.220) | -0.90 (1.810)

10. Secondary Outcome: Change From Baseline in Hirsutism at Week 28 Using the Ferriman-Gallwey Score (Females Only) at Week 28
Description: Ferriman-Gallwey score is a method used to assess and quantify hirsutism in women. A total score < 8 is considered normal whereas a score of 8 to 15 indicates mild hirsutism. A score >15 indicates moderate or severe hirsutism. The Ferriman-Gallwey score ranged from 0 to 36. Higher score indicated more hirsutism. Change from baseline is reported (negative change from baseline indicated improvement).
  LS mean was assessed using ANCOVA. Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline, Week 28
Population: FAS: All participants with CAH who were randomized into the study and who received at least 1 dose of study drug. Only female participants with evaluable data for the endpoint were analyzed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 16 | 13
score on a scale | -1.0 [-2.5 to 0.6] | -1.2 [-3.0 to 0.5]

11. Secondary Outcome: Change From Baseline in Acne Using the Global Evaluation Acne (GEA) Scale (Females Only) at Week 28
Description: Acne severity was assessed according to GEA scale, which ranged from 0 (Clear. No lesions) to 5 (Very severe). Higher score indicated higher severity of acne. Change from baseline is reported (negative change from baseline indicated improvement).
  LS mean was assessed using ANCOVA. Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline, Week 28
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 16 | 13
score on a scale | -0.3 [-0.5 to -0.1] | -0.2 [-0.4 to 0.0]

12. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) Percent Levels at Week 28
Description: LS mean was assessed by ANCOVA. Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline, Week 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent HbA1c
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 22 | 24
percent HbA1c | -0.01 [-0.09 to 0.06] | -0.06 [-0.13 to 0.01]

13. Secondary Outcome: Change From Baseline in Waist Circumference at Week 28
Description: as for outcome 6
Time Frame: Baseline, Week 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 24 | 24
centimeters | 0.867 [-1.387 to 3.121] | -1.242 [-3.496 to 1.012]

14. Secondary Outcome: Change From Baseline in Body Weight at Week 28
Description: as for outcome 12
Time Frame: Baseline, Week 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 25 | 25
kilograms | 1.29 [0.00 to 2.58] | -1.67 [-2.96 to -0.38]

15. Secondary Outcome: Change From Baseline Quality of Life Using the Self-completed Medical Outcome Study 36-Item Short Form Health Survey (SF-36) Total Score for the Physical and Mental Components and the Sub-domain of Vitality at Week 28
Description: SF-36 evaluates aspects of functional health and well-being. The physical component has 4 sub-scales: physical function, role limitations due to physical problems, pain, and general health perception; and the mental component has 4 sub-scales: vitality, social function, role limitations due to emotional problems, and mental health. Total scores for the physical and mental component are presented as well as the sub-scale score for vitality. Scores were summarized and transformed into a range from 0 to 100; 0=worst, and 100=best outcome. Higher scores indicated better outcome. Change from baseline is reported (positive change from baseline indicated improvement).
  LS mean was assessed by ANCOVA. Assessment of efficacy at Week 28 was a composite of each participant's on-treatment visit closest in time to 28 weeks post randomization.
Time Frame: Baseline, Week 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Chronocort | Cortef
Number analyzed (Participants) | 21 | 15
score on a scale
  Physical Component | -3.313 [-5.801 to -0.824] | -1.031 [-3.976 to 1.913]
  Mental Component | 0.772 [-3.209 to 4.752] | 0.685 [-4.034 to 5.403]
  Vitality Sub-domain | -0.847 [-4.354 to 2.660] | -0.002 [-4.157 to 4.153]

ADVERSE EVENTS:
Time Frame: Up to 30 days after last study dose (maximum treatment duration of approximately 53 weeks; median exposure = 255.0 days for Chronocort and 230.5 days for Cortef)
Description: The Cortef Run-in reporting group was assessed using the screening population. The Cortef and Chronocort reporting groups were assessed using the safety analysis set that included all participants who were randomized and received at least 1 dose of study drug in the treatment period.
Groups:
- Cortef Run-In: Participants received Cortef 30 mg total daily dose during the run-in therapy for 4 weeks prior to randomization.
Arm/Group | Cortef Run-In | Chronocort | Cortef
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/55 | 2/25 | 1/28
Other Adverse Events (participants affected / at risk) | 2/55 | 22/25 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cortef Run-In (N=55) | Chronocort (N=25) | Cortef (N=28)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cortef Run-In (N=55) | Chronocort (N=25) | Cortef (N=28)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 4 (6) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 6 (6)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Weight increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 3 (4)
Stress (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT05063994/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT05063994/SAP_001.pdf